CLINICAL TRIAL: NCT05421026
Title: Cyberbullying Among Sohag University Students , Egypt .
Brief Title: Cyberbullying Among Sohag University Student
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amera Fayez Shenouda, Demonstrator at public health and community department at Sohag University, Sohag University
Other Study IDs: Soh-Med-22-06-01
Record Dates: First submitted 2022-06-12; First posted 2022-06-16 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Cyberbullying Among Sohag University Students
Keywords: cyberbullying
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cyberbullying can be defined as intentional aggression through electronic routes, such as text messages, e-mails, chat rooms, online games, and social websites. In comparison with traditional bullying, cyberbullying has many unique characteristics that boost its harmful effects, including the inability to avoid bullying, presence of larger and more potential audience, the continuity of bullying regardless of time or place, and the anonymity of perpetrator in many occasions .

DETAILED DESCRIPTION:
In Egypt almost half of Beni-sueif university students (48.2%) reported experiencing cyberbullying victimization. Female students, students living in urban areas and those who spent more hours using the internet reported more exposure (p<0.001). Harassment was the main type stated by females (79.8%) while flaming was excessively reported by males (51.8%). Students responded mostly by anger (63.1%), hatred (23.2%) and sorrow (22.6%) towards the worst victimization incidents.

In this study I want to study the situation of cyberbullying among Sohag University students .

, study patterns of cyberbullying among Sohag University students , determine of correlates of cyberbullying among Sohag University students such as family factors and study the implications of cyberbullying on victims .

ELIGIBILITY:
Inclusion Criteria:

* students of the selected faculties

Exclusion Criteria:

* students who will refuse to participate in this study.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample was taken by the mean of cluster random sampling technique among all sohag faculties. Four faculties were chosen; Two practical faculties and two theoritical faculties . Then a suitable random sample will be taken from the students of the determined faculties.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
study the situation of cyberbullying among Sohag University students | 2022-2023
  study the prevalence , the pattern and correlates of cyberbullying